CLINICAL TRIAL: NCT06056687
Title: Effect of Alpha-lipoic Acid on Inflammatory and Cardiac Fibrosis Markers in Diabetic Patients With Ischemic Cardiomyopathy
Brief Title: Alpha-lipoic Acid in Diabetic Patients With Ischemic Cardiomyopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Associate Professor, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALA in Ischemic Cardiomyopathy
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Ischemic Cardiomyopathy; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Thioctic Acid; Tablets

STUDY DESIGN:
Intervention Model Description: 60 patients with type II Diabetes Mellitus with Ischemic Cardiomyopathy on optimal standard medical therapy, who will be consecutively randomized into two groups, group on ALA 600 mg once daily and the second group on placebo.
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alpha Lipoic Acid Group (Experimental): ALA 600 mg once daily
  Interventions: Drug: Alpha Lipoic Acid 600 MG Oral Tablet
- Placebo Group (Placebo Comparator): the second group on placebo once daily
  Interventions: Other: Placebo Tablet

INTERVENTIONS:
Drug: Alpha Lipoic Acid 600 MG Oral Tablet — Alpha Lipoic Acid 600 MG Oral Tablet once daily
  Other Names: Thiotacid 600 mg
  Arms: Alpha Lipoic Acid Group
Other: Placebo Tablet — Placebo Tablet once daily
  Other Names: Placebo
  Arms: Placebo Group

SUMMARY:
The aim of this study is to investigate the effect of alpha-lipoic acid on inflammatory markers and cardiac fibrosis markers in diabetic patients with Ischemic Cardiomyopathy.

DETAILED DESCRIPTION:
* A 3-month, prospective double blind interventional study, which will include 60 patients with type II Diabetes Mellitus with Ischemic Cardiomyopathy on optimal standard medical therapy, who will be consecutively randomized into two groups, group on ALA 600 mg once daily and the second group on placebo once daily.
* Approval will be obtained from Research and Ethics Committee of Faculty of Pharmacy, Damanhour University. A written informed consent will be obtained from patients before begining of the study.
* All patients will undergo complete physical examination at baseline and after 3 months of treatment.
* Patients will be assessed using Echocardiography before and after the study focusing on:

Left atrial diameter (LAD), basic left ventricular dimensions (EDD and ESD) and both systolic and diastolic function.

-Measurements of inflammatory markers such as [C-reactive protein (CRP), Tumor necrosis factor alpha (TNFα)] and fibrosis markers such as [Transforming growth factor beta (TGFβ), Matrix metalloproteinase 2 (MMP-2)] at the beginning of the study and after 3 months of the study.

Study Outcomes: all patients will be followed up for 3 months for:

* 1ry outcomes: Change in inflammatory and fibrosis markers levels. LV Echocardiography improvements of any of basic Echo parameters.
* 2ry outcomes: Major Adverse Cardiovascular Events (MACE) such as MI, stroke or death. any side effects of the drug. Results The results of the study will be tabulated and statistical tests appropriate to the study will be conducted to evaluate significance of results.

conclusion Conclusion, and recommendations will be given.

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes with a history of CAD.
* LV ejection fraction (LVEF) ≤40%.
* Ischemic heart failure patients with NYHA grade II-IV.

Exclusion criteria:

* Type 1 diabetes.
* Severe CKD with GFR ≤ 15 ml/min/1.73m^2.
* Severe liver disease.
* Thyroid disorders.
* Acute febrile illness.
* Autoimmune disorders or connective tissue disorders.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
C-reactive protein (CRP) | 3 month
  Serum Biomarker (mg/ml)
Tumor necrosis factor alpha (TNFα)] | 3 Months
  Serum Biomarker (pg/ml)
Transforming growth factor beta (TGFβ) | 3 Months
  fibrosis markers (ng/ml)
Matrix metalloproteinase 2 (MMP-2) | 3 Months
  fibrosis markers (ng/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Ass Prof., Study Chair — Damanhour University; Noha El bassiouny, Lecturer, Study Director — Damanhour University
Locations (1):
- Damanhour Teaching Hospital, General Organization for Teaching Hospitals and Institutes., Damanhūr, Elbehairah, Egypt